CLINICAL TRIAL: NCT03357991
Title: Performance of E6/E7 mRNA to Detect Anal High-Grade Intraepithelial Lesions and Cost-effectiveness Analysis of a New Screening Strategy for Anal Cancer in HIV Positive Men Who Have Sex With Men
Brief Title: E6/E7 mRNA Performance to Detect HSIL and Cost-effectiveness Analysis of This Screening Strategy in HIV + MSM
Acronym: ELAVI-67
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Universitari de Bellvitge (Other)
Collaborators: Institut d'Investigació Biomèdica de Bellvitge (Other)
Responsible Party: Principal Investigator, Daniel Podzamczer Palter, PhD. Chief of the HIV and STD Unit (Infectious Disease Service), Hospital Universitari de Bellvitge
Other Study IDs: PR076/17; PI16/01056 (Other Grant/Funding Number: Instituto de Salud Carlos III)
Record Dates: First submitted 2017-11-24; First posted 2017-11-30 (Actual); Last update posted 2017-12-07 (Actual); Status verified 2017-12

CONDITIONS: HPV - Anogenital Human Papilloma Virus Infection; HSIL, High Grade Squamous Intraepithelial Lesions; Anal Cancer; Hiv
Keywords: E6/E7 mRNA; anal cancer screening; men who have sex with men; cost-effectiveness analysis; High resolution anoscopy
MeSH Terms: conditions — Squamous Intraepithelial Lesions; Anus Neoplasms; Acquired Immunodeficiency Syndrome; Homosexuality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — 1. Detection of anal HPV
     * Hybrid Capture® 2 HPV DNA (QIAGEN Inc., Gaithersburg, Maryland; EE.UU): enzyme linked immunoabsorvent assay based on a sandwich hybridisation that allows a qualitative measure of DNA of 13 HPV.
     * Linear Array HPV Genotyping Test (Roche Molecular Systems Inc., Alameda, California, EE.UU): it detects a region within the HPV L1 that share 37 anogenital HPV genotypes.
     * Detection of E6/E7 VPH mRNA using APTIMA® HPV Test (Gen-Probe Inc., San Diego, California, EE.UU): it allows the qualitative detection of HPV E6/E7 mRNA from 14 high-risk HPVs.
  2. Anal cytology: processed with Thinprep Pap Test (Hologic, Marlborough, Massachusetts, USA). The swab is deposited into preserved liquid based cytology: PreservCyt Solution.
  3. HRA with biopsy of suspicious lesions
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study evaluates the positive and negative predictive value of E6/E7 mRNA expression for anal HSIL and its capacity to predict incident HSIL in HIV + MSM. We also analyse the cost-effectiveness of this new screening strategy. It is an ambispective study with 355 participants and a follow-up period of 2 to 5 years.

DETAILED DESCRIPTION:
Introduction: Anal cancer incidence is increasing in HIV-infected men who have sex with men (MSM). There are still no standardized criteria for anal cancer screening. Anal cytology has not shown enough sensitivity and specificity in the selection of patients who need more invasive procedures, as high resolution anoscopy (HRA). Human Papillomavirus (HPV) E6 and E7 oncogenes deregulation is a crucial factor in neoplasic lesions progression.

Objectives: 1)To assess the negative and positive predictive value of E6/E7 mRNA expression for high-grade squamous intraepithelial lesions (HSIL) and its capacity to predict the incidence of new HSIL during the follow-up 2)To analyze the cost-effectiveness of E6/E7 as a new screening strategy for anal cancer compared with usual strategies (cytology and DNA detection).

Methodology: Ambispective longitudinal study. Participants: HIV MSM from the outpatients HIV and STD Unit of Bellvitge Hospital. We include patients visited within the usual outpatient practice since January 2015 with a cytology stored following the Hospital protocol, as well as patients collected prospectively since January 2017. This methodological approach will let to reduce the time of inclusion and maximize follow-up time. Sample size calculated: 355 participants. Follow-up period: 2 to 5 years. At each visit an anal smear for cytology, HPV DNA detection (by Linear Array and Hybrid Capture) and E6/E7 mRNA expression and a HRA with biopsy of suspicious areas of dysplasia will be performed. The analysis of cost-effectiveness will be made with a Markov model that projects long-term cost and effectiveness for both strategies, the E6/E7 and conventional cytology plus detection of High Risk HPV.

ELIGIBILITY:
Inclusion Criteria:

* Men who have sex with men >= 18 years
* HIV documented infection
* Signature of the informed consent

Exclusion Criteria:

* Previous diagnosis of anal cancer.
* Treatment of anal intraepithelial lesions the 5 years before study inclusion.
* Suspect infiltrating anal cancer, requiring exploration under anesthesia and surgical removal for histological confirmation.
* History of diffuse ano-genital condylomatous disease the 5 years before study inclusion or presence at first visit.
* Other factors that could prevent correct diagnosis and monitoring of the anal dysplastic lesions (test intolerance, proctological pathology that does not allow HRA, etc.).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult HIV-infected MSM visited in the HIV Unit of Bellvitge's University Hospital and underwent routine anal cancer screening.
  Retrospective participants: patients attended between January 2015 and December 2016 and with part of the anal smear sample stored.
  Prospective participants: patients who start anal cancer screening during the inclusion period.
Sampling Method: Probability Sample
Enrollment: 355 (Estimated)
Dates: Start 2015-01-11 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Determine the predictive value of HPV E6/E7 mRNA for the detection of HSIL and its ability to predict incident cases. | 2-5 years
  Determination of HPV E6/E7 ARNm in anal samples of 355 HIV + MSM. Correlation of the detection of HPV E6/E7 ARNm with the diagnosis of HSIL in this patients performing anal cytology an HRA at the first visit and during the follow-up.

SECONDARY OUTCOMES:
Cost-effectiveness analysis of an anal cancer screening strategy based on HPV E6/E7 mRNA analysis. | 2-5 years
  Cost-effectiveness analysis of an anal cancer screening strategy based on the selection of candidates for HRA according to the expression of the E6 / E7 mRNA, compared to the usual strategy based on cytology and DNA HPV detection.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Podzamczer Palter, Principal Investigator — Hospital Universitari de Bellvitge
Locations (1):
- Hospital Universitary de bellvitge, L'Hospitalet de Llobregat, Barcelona, Spain

REFERENCES:
- [Derived] Torres M, Silva-Klug A, Ferrer E, Saumoy M, Trenti L, Tous S, Esteban A, Baixeras N, Catala I, Vidal A, G Bravo I, Podzamczer D, de Sanjose S. Detecting anal human papillomavirus infection in men who have sex with men living with HIV: implications of assay variability. Sex Transm Infect. 2023 May;99(3):187-190. doi: 10.1136/sextrans-2021-055303. Epub 2022 May 11. PMID 35545433